CLINICAL TRIAL: NCT07234253
Title: Developing and Evaluating a Culturally Sensitive Sexual Health Education Program for Autistic Young Adults in South Korea With Input From a Community Advisory Board
Brief Title: Sexuality and Relationship Education Program for Autistic Young Adults in South Korea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: National Research Foundation of Korea (Other); Korean Association for Persons with Autism (Unknown); Smile Together Foundation (Unknown)
Responsible Party: Principal Investigator, So Hyun Kim, Associate Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-0055-10
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Autistic young adults will receive a group-based sexuality and relationship education program delivered in a telehealth format over 10 sessions (90 minutes per session, once a week for 10 weeks). The program will cover the following topics: social relationship (e.g., distinguishing types of relationships, apologizing, and refusing), romantic relationships, consent, sexual behavior, reproduction, prevention of sexual harassment, online and social media use related to sexuality, gender, and sexual orientation.
  Interventions: Behavioral: Our Love, Our Style (OLOS)

INTERVENTIONS:
Behavioral: Our Love, Our Style (OLOS) — The intervention will consist of an online, group-based sexuality and relationship education program delivered over 10 sessions (90 minutes per session, once a week for 10 weeks). The program will cover the following topics, adapted to the Korean cultural context and the needs of autistic young adults aged 18-35 years: social relationships (e.g., distinguishing types of relationships, apologizing, and refusing), romantic relationships, consent, sexual behavior, reproduction, prevention of sexual harassment, online and social media use related to sexuality, gender, and sexual orientation.

SUMMARY:
The goal of this single-arm clinical trial is to conduct a preliminary evaluation of Our Love, Our Style, a group-based sexuality and relationship education program for autistic young adults in South Korea. The study aims to examine the preliminary efficacy of the program by assessing increases in sexuality knowledge, sexual and relationship behaviors, and motivation. It will also evaluate the feasibility and acceptability of implementing the program among Korean autistic young adults.

Participants will receive a 10-session, online, group-based program (90 minutes per session, once a week for 10 weeks) delivered via telehealth. The program is adapted to the Korean cultural context and tailored to the needs of autistic young adults aged 18-35 years. It will cover the following topics: social relationships (e.g., distinguishing types of relationships, apologizing, and refusing), romantic relationships, consent, sexual behavior, reproduction, prevention of sexual harassment, online and social media use related to sexuality, gender, and sexual orientation.

ELIGIBILITY:
Inclusion Criteria:

* previous medical diagnosis of autism spectrum disorder (ASD) or ASD based on DSM-5 using Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
* Verbal ability sufficient to produce full sentences (i.e. ADOS-2 Module 4 language level)
* Full-Scale IQ equal to or above 70

Exclusion Criteria:

- Presence of prominent hallucinations or delusions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Psychosexual Knowledge Test (PKT) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 37-item multiple-choice test designed to assess a broad range of psychosexual knowledge, from understanding physical terminology to applied sexual and psychological concepts. Each item is scored as True/False
Perceived Knowledge Questionnaire (PKQ) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 5-item self-report measure evaluating participants' perceived level of sexual health knowledge. Items are answered in a True/False format.
Korean Relationship and Sexuality Scale (KRSS) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 150-item self-report scale developed to comprehensively evaluate sexual health knowledge and understanding of relationships, corresponding to the content covered in the intervention program. Visual aids are provided to support autistic participants' comfort with visual materials. Each item is rated as Agree or Disagree.
Sexual Desire Inventory-2 (SDI-2) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 14-item self-report questionnaire measuring the frequency and intensity of sexual desire across various contexts. Items are rated on an 8-point scale ranging from 0 (Not at all) to 7 (More than once a day).
Self-Efficacy in Romantic Relationships Scale | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 12-item scale assessing self-efficacy and beliefs regarding one's ability to maintain and manage romantic relationships. Each item is rated on a 9-point Likert scale from 1 (Strongly disagree) to 9 (Strongly agree).
Sexual and Dating Experiences Questionnaire | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 7-item multiple-choice questionnaire evaluating participants' experiences with various intimate and dating behaviors. Each item is answered as Never, Once or twice, or More than twice.
Sexual Experience Questionnaire (SEQ) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention (follow-up).
  A 12-item instrument assessing the frequency of diverse sexual experiences. Responses are recorded using a four-point frequency scale: Never, Once, A few times, or Many times.
Program Feasibility Survey | post-intervention (1 week after the completion of the intervention)
  This questionnaire will be completed by participants at the end of the intervention program to assess the feasibility of the intervention. It includes items evaluating the practicality and usability of the program (e.g., "The online platform was easy to use," "I was able to find time to complete assigned tasks"). Each item is rated on a 5-point Likert scale (1 = strongly disagree, 3 = neutral, 5 = strongly agree). Scores for each item range from 1 to 5, with higher scores indicating that participants perceived the program as more feasible.
Program Acceptability Survey | post-intervention (1 week after the completion of the intervention)
  This questionnaire will be completed by participants at the end of the intervention program to assess the acceptability and overall satisfaction with the intervention. It includes items evaluating perceived benefits of the sessions (e.g., "I benefited from the sessions with the interventionist"). Each item is rated on a 5-point Likert scale (1 = strongly disagree, 3 = neutral, 5 = strongly agree). Scores for each item range from 1 to 5, with higher scores indicating that participants perceived the program as more acceptable.

SECONDARY OUTCOMES:
Camouflaging Autistic Traits Questionnaire (CAT-Q) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  A 25-item self-report questionnaire assessing social camouflaging behaviors used to mask autistic traits. It includes three subscales: Compensation, Masking, and Assimilation.Items are rated on a 7-point Likert scale, and the measure includes reverse-scored items. Total scores range from 25 to 175, with higher scores indicating greater use of camouflaging behaviors. The Compensation subscale ranges from 9 to 63 points, and the Masking and Assimilation subscales each range from 8 to 56 points, with higher scores reflecting more frequent use of the respective camouflaging strategies.
Korean-Adolescents/Adults Sensory Profile (K-AASP) | Baseline (pre-intervention)
  A 60-item self-report measure assessing behavioral responses to everyday sensory experiences among individuals aged 11-65 years. Each item is rated on a 5-point scale from Almost never to Almost always.
Beck Depression Inventory (BDI) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  A 21-item self-report instrument measuring the severity of depressive symptoms experienced during the past week. Each item is rated on a 0-3 scale, yielding a total score range of 0-63. Higher scores indicate more severe depressive symptoms.
Beck Anxiety Inventory (BAI) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  A 21-item self-report instrument assessing the severity of anxiety symptoms, including cognitive, emotional, and physiological aspects of anxiety and panic. Each item is rated on a 0-3 scale, yielding a total score range of 0-63. Higher scores indicate more severe anxiety symptoms.
UCLA Loneliness Scale (Korean Short Form) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  An 8-item short form of the UCLA Loneliness Scale assessing perceived loneliness using a 4-point Likert scale (1 = Never to 4 = Often). Higher scores indicate greater loneliness.
Loneliness and Social Isolation Scale | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  A 6-item self-report measure assessing both objective and subjective dimensions of social isolation, including social networks, perceived social support, and loneliness. Each item is rated from 0 to 3.
Discrimination and Stigma Scale (DISC-12) | Baseline (pre-intervention)
  A 34-item measure assessing experiences of stigma and discrimination related to mental health issues. It includes four subdomains: unfair treatment, self-limiting behavior, coping with stigma, and positive discrimination. Each item is rated on a 4-point scale from Not at all to A lot.
Relationships, Employment, Autonomy, and Life Satisfaction Scale (REALS) | Baseline (pre-intervention), 1 week post-intervention, and 10 weeks post-intervention follow-up.
  A self-report measure developed for adults with autism or other intellectual and developmental disabilities. It assesses 19 life domains-including relationships, employment, autonomy, daily living, and satisfaction-using ratings of frequency, support, and satisfaction. The REALS provides several types of response options. Frequency items, used when the key question concerns how often a person engages in a particular behavior, are rated on a 5-point scale from 0 (never) to 4 (often), with higher scores indicating more frequent engagement. Support items, used to understand the level of assistance needed in a domain or the degree to which an individual can perform tasks independently, are rated from 0 to 4, where higher scores indicate greater independence and less need for support. Satisfaction items, which assess how satisfied an individual is with various aspects of their life, are rated on a 0-3 scale, with higher scores reflecting greater satisfaction in that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Boin Choi, PhD, Study Director — Ewha Womans University
Locations (1):
- Korea University, Seoul, South Korea